CLINICAL TRIAL: NCT00834886
Title: Delayed Sleep Phase Syndrome in Adolescents and Young Adults. Sleep, Personality, Developmental History, Circadian Rhythm, Daytime Functioning and Treatment
Brief Title: Randomized Controlled Trial on the Treatment Effects of Melatonin and Light Therapy on Delayed Sleep Phase Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Bjorn Bjorvatn, Professor, MD, PhD, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00834886
Record Dates: First submitted 2009-01-09; First posted 2009-02-03 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Delayed Sleep Phase Syndrome
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Combination (Active Comparator): Bright light 10.000 lux + melatonin 3 mg
  Interventions: Dietary Supplement: Melatonin; Other: Bright light
- Melatonin (Active Comparator): Melatonin 3 mg + placebo red light 400 lux
  Interventions: Dietary Supplement: Melatonin; Other: Placebo red light
- Bright light (Active Comparator): Bright light 10.000 lux + placebo capsule 3 mg rice flour
  Interventions: Other: Bright light; Other: Placebo capsule
- Placebo (Placebo Comparator): Placebo Red light 400 lux + placebo capsule 3 mg rice flour
  Interventions: Other: Placebo red light; Other: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Melatonin — Capsules, 3 mg, once every night
  Other Names: Nature´s One melatonin, by Asman, Inc.
  Arms: Combination; Melatonin
Other: Bright light — Bright light therapy 10.000 lux by Miljølys AS
  Arms: Bright light; Combination
Other: Placebo red light — Red light 400 lux as placebo light
  Arms: Melatonin; Placebo
Other: Placebo capsule — Capsules containing 3 mng rice flour, once every night
  Arms: Bright light; Placebo

SUMMARY:
In this study the investigators will examine the effects of melatonin and light therapy on delayed sleep phase syndrome in adolescents 16 up to 20 years old. 60 subjects will be randomized into four different groups; melatonin + light therapy (N=15), melatonin + placebo light (N=15), placebo + light therapy (N=15) and placebo + placebo light. This is a double-blinded treatment and the participants will receive this treatment for 2 weeks. Then they will be re-randomized into two groups; full treatment with light therapy + melatonin (N=30) and no treatment (N=30) for 3 months unblinded. The investigators will test the subjects pre-treatment, post 2 week treatment and after 3 months.

DETAILED DESCRIPTION:
Delayed sleep phase syndrome (DSPS) is a circadian rhythm sleep disorder where the sleep-wake rhythm is significantly delayed according to the environmental demands. Hence, the symptoms consist of major difficulties falling asleep and problems awakening in due time and patients often experience work- and school related impairments (The International Classification of Sleep Disorders: Diagnostic and Coding manual, 2005). However, correct diagnosis is often not made and the treatment offered is, accordingly, often inadequate. DSPS normally develops in interplay between dysfunctional habits/behaviour and biological vulnerability.

Bright light therapy and administration of exogenous melatonin comprise the most common interventions. Timed bright light has been shown to effectively phase advance the rhythm (Rosenthal et al., 1990), but no standardized guidelines regarding the duration, intensity or timing of light exposure have been established. Compliance to the treatment is often poor because it involves structuring the daily schedule, which may be hard for the relevant age group. Similarly, administration of melatonin in the evening has been shown to phase advance the rhythm (Lewy et al., 1998; Mundey, Benloucif, Harsanyi, Dubocovich, & Zee, 2005), but a standardized approach for dose, duration and timing is lacking.

It is important to establish effective treatment guidelines for delayed sleep phase syndrome. Large scale studies on the effects of melatonin and bright light treatment in randomized placebo-controlled designs are needed. In a clinical trial we aim to investigate the efficacy of bright light and melatonin treatment using a 4 armed randomized placebo controlled design.

ELIGIBILITY:
Inclusion Criteria:

* 16-25 years old
* lives in the Bergen area
* has Delayed Sleep Phase Disorder

Exclusion Criteria:

* pregnant or nursing women
* other sleep disorders (i.e. sleep apnoea or PLMS)
* moderate to serious psychiatric disease
* use of psychopharmacological medicines
* in psychotherapeutic treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Bjorvatn, MD., PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Publications from the stury are reported here. IPD can be retrieved upon request to the study investigator.

REFERENCES:
- [Result] Wilhelmsen-Langeland A, Saxvig IW, Pallesen S, Nordhus IH, Vedaa O, Lundervold AJ, Bjorvatn B. A randomized controlled trial with bright light and melatonin for the treatment of delayed sleep phase disorder: effects on subjective and objective sleepiness and cognitive function. J Biol Rhythms. 2013 Oct;28(5):306-21. doi: 10.1177/0748730413500126. PMID 24132057
- [Result] Saxvig IW, Wilhelmsen-Langeland A, Pallesen S, Vedaa O, Nordhus IH, Bjorvatn B. A randomized controlled trial with bright light and melatonin for delayed sleep phase disorder: effects on subjective and objective sleep. Chronobiol Int. 2014 Feb;31(1):72-86. doi: 10.3109/07420528.2013.823200. Epub 2013 Oct 21. PMID 24144243

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination: Melatonin: Capsules, 3 mg, once every night
  Light therapy: Light therapy 10.000 lux by Miljølys AS
- Melatonin: Melatonin: Capsules, 3 mg, once every night
  placebo light therapy: Placebo light
- Bright Light: Placebo melatonin: Capsule 3 mg, rice flour
  Light therapy: Light therapy 10.000 lux by Miljølys AS
- Placebo: Placebo melatonin + placebo light therapy
  Placebo melatonin: Capsule 3 mg, rice flour
  placebo light therapy: Placebo light
Period: Overall Study
Arm/Group | Combination | Melatonin | Bright Light | Placebo
Started | 10 | 10 | 10 | 10
Completed | 10 | 9 | 9 | 10
Not Completed | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Melatonin and Light Therapy: Melatonin: Capsules, 3 mg, once every night
  Light therapy: Light therapy 10.000 lux by Miljølys AS
- Melatonin and Placebo Light: Melatonin: Capsules, 3 mg, once every night
  placebo light therapy: Placebo light
- Placebo Melatonin and Light Therapy: Placebo melatonin: Capsule 3 mg, rice flour
  Light therapy: Light therapy 10.000 lux by Miljølys AS
- Placebo Melatonin and Placebo Light: Placebo melatonin + placebo light therapy
  Placebo melatonin: Capsule 3 mg, rice flour
  placebo light therapy: Placebo light
- Total: Total of all reporting groups
Arm/Group | Melatonin and Light Therapy | Melatonin and Placebo Light | Placebo Melatonin and Light Therapy | Placebo Melatonin and Placebo Light | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 20.3 (3.3) | 21.2 (2.7) | 20.7 (3.4) | 20.8 (3.4) | 20.7 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 8 | 7 | 28
  Male | 2 | 5 | 2 | 3 | 12
Region of Enrollment [Number; unit: participants]
  Norway | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: To Investigate the Efficacy on Rise Time of Bright Light Therapy and Melatonin Treatment Using a 4 Armed Placebo Controlled Design. Main Outcome Measures: Sleep Log, Actigraphy and Psychological Tests.
Description: Sleep diary, rise time (when participants rise from bed in the morning, self-report) before and after a randomized controlled 4 armed treatment study including a follow-up 3 months later.
  Midnight is 0000; in the outcome measure table the value is given in minutes after midnight.
  i.e. 530 equals 08:50 in the morning.
Time Frame: 1 day after two-week treatment ends
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Combination: Bright light + melatonin
  Melatonin: Capsules, 3 mg, once every night
  Light therapy: Light therapy 10.000 lux by Miljølys AS
- Melatonin: Melatonin + placebo light
  Melatonin: Capsules, 3 mg, once every night
  placebo light therapy: Placebo light
- Bright Light: Bright light + placebo capsule
  Placebo melatonin: Capsule 3 mg, rice flour
  Light therapy: Light therapy 10.000 lux by Miljølys AS
- Placebo: Placebo capsule + placebo light
  Placebo melatonin: Capsule 3 mg, rice flour
  placebo light therapy: Placebo light
Arm/Group | Combination | Melatonin | Bright Light | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Minutes | 530 (121) | 506 (98) | 520 (148) | 543 (163)

2. Primary Outcome: To Investigate the Efficacy on Subjective Sleepiness of Bright Light Therapy and Melatonin Treatment Using a 4 Armed Placebo Controlled Design. Main Outcome Measures: Sleep Log, Actigraphy and Psychological Tests.
Description: Subjective sleepiness; Karolinska sleepiness scale (KSS). The KSS is a scale in which the subjects rate their concurrent sleepiness level. The scale is verbally anchored with steps ranging from 1 ("very alert") to 9 ("very sleepy, fighting sleep, effort to stay awake").
Time Frame: 1 day after 2-week treatment ended
Population: All participants in the four arms
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combination | Melatonin | Bright Light | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale | 6.0 (1.6) | 5.9 (1.3) | 6.3 (1.8) | 6.5 (1.5)

3. Primary Outcome: To Investigate the Efficacy on Sleep Onsel Latency of Bright Light Therapy and Melatonin Treatment Using a 4 Armed Placebo Controlled Design. Main Outcome Measures: Sleep Log, Actigraphy and Psychological Tests.
Description: Actigraphy, sleep onset latency (SOL). An actigraph is a wrist-worn movement sensor that objectively record motor activity. Participants used an event button to mark bed time and rise time. The actiwatch is waterproof and participants were instructed not to take it off at any time during the data collection peroid.
Time Frame: 1 day after 2-week treatment ended
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Combination | Melatonin | Bright Light | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Minutes | 11 (8) | 21 (19) | 15 (10) | 24 (11)

ADVERSE EVENTS:
Arm/Group | Combination | Melatonin | Bright Light | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 4/10 | 3/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination (N=10) | Melatonin (N=10) | Bright Light (N=10) | Placebo (N=10)
Headache (Nervous system disorders) | 2 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Discomfort in eyes (Eye disorders) | 2 | 1 | 1 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No